CLINICAL TRIAL: NCT02007317
Title: A Single Center, Open Label Study for Evaluation of the Safety and Efficacy of Oshadi D and Oshadi R in Patients With Basal Cell Carcinoma (BCC) Prior to Tumor Excision- a Phase II Study
Brief Title: Safety and Efficacy of Oshadi D and Oshadi R in Basal Cell Carcinoma Patients Prior to Tumor Excision a Phase 2 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-BCC-P2-01
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2016-03

CONDITIONS: BCC
Keywords: BCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi D and Oshadi R (Experimental): Anti tumor agents
  Interventions: Drug: Oshadi D & Oshadi R

INTERVENTIONS:
Drug: Oshadi D & Oshadi R — Anti tumor agents

SUMMARY:
This study is single-arm, none randomized, open label, two-dose-cohorts, single center clinical trial for evaluation of the safety and efficacy of Oshadi D and Oshadi R in patients with BCC. Patients will receive Oshadi D and Oshadi R for 60 -90 days until the planned surgical excision of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years old with tissue confirmed diagnosis of local BCC.
* Patient is candidate for surgical excision of the BCC in few months.
* BCC lesion ≥10mm in its longest diameter.
* Sexually active fertile patients and their partners must agree to use medically accepted methods of contraception during therapy and 3 months after the last dose of the study drugs.
* Female patients of childbearing potential must have a negative pregnancy test at screening.
* Patient must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.

Exclusion Criteria:

* Uncontrolled Intercurrent illness or any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Other active cancer disease.
* Serum creatinine > 1.5 mg/dL for males and >1.4 mg/dL for females.
* Female patient who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Any acute cardiovascular event during the last 6 months prior to inclusion.
* Symptomatic congestive heart failure with ejection fraction < 30%.
* Patient has prothrombin time/International Normalization Ration (PT/INR) or partial thromboplastin time (PTT) test results > 1.3 UNL.
* Hemoglobin ≤ 11 g/dL
* Platelets < 150,000 per microliter
* White blood cell count<3,000 x109/L and/or absolute neutrophils count <1.5 x 109/L
* Significant swallowing disorders.
* History of small bowel surgery.
* Any history of pelvic or abdominal radiation.
* Pre-existing mal-absorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption.
* Mental disorders.
* Inability to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurence | treatment end (day 60 or 90)

SECONDARY OUTCOMES:
The primary efficacy endpoint of this study is Overall Response Rate (ORR) | treatment end (day 60 or 90)

OTHER OUTCOMES:
To estimate the duration of treatment to achieve response | 9 months
  To estimate the duration of treatment needed to achieve response

CONTACTS AND LOCATIONS:
Overall Officials: Lior Heller, Prof., Principal Investigator — Assaf Harofeh Medical Center, Zrifin, Israel
Locations (1):
- Assaf-Harofeh Medical Center, Zrifin, Israel